CLINICAL TRIAL: NCT04839510
Title: An Open-label, Single-arm, Multi-center, Phase II Clinical Study of MRG002 in the Treatment of Patients With HER2-positive Unresectable Locally Advanced or Metastatic Urothelium Cancer
Brief Title: A Study of MRG002 in the Treatment of HER2-positive Unresectable Locally Advanced or Metastatic Urothelium Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG002-006
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Locally Advanced Urothelial Cancer; Metastatic Urothelial Carcinoma
Keywords: MRG002; Antibody Drug Conjugate (ADC); HER2; Urothelium Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG002 (Experimental): MRG002 will be administrated by an IV infusion of 2.6 mg/kg on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG002

INTERVENTIONS:
Drug: MRG002 — Administrated intravenously

SUMMARY:
The objective of this study is to assess the safety, efficacy, pharmacokinetics, and immunogenicity of MRG002 as single agent in patients with HER2-positive unresectable locally advanced or metastatic urothelium cancer.

DETAILED DESCRIPTION:
The study consists of two stages. In Phase IIa, approximately 25 subjects will be enrolled to evaluate the safety and preliminarily efficacy of MRG002. Based on the initial safety and efficacy data obtained from the Phase IIa, the study design of second stage Phase IIb single-arm study either will be continued or the trail will be terminated. If the Phase IIa data support the continuation of the study, in the second stage, approximately an additional 33 subjects will be enrolled to further evaluate the efficacy and safety of MRG002.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the ICF and follow the requirements specified in the protocol.
2. Aged 18 to 75 (including 18 and 75), both genders.
3. Expected survival time ≥ 12 weeks.
4. Patients with unresectable locally advanced or metastatic urothelium cancer confirmed by histopathology.
5. Failed in the prior one or more line of systemic chemotherapy.
6. HER2 positive (IHC 3 + or IHC 2 +) in the tumor specimens confirmed by central laboratory test.
7. Archival or biopsy tumor specimens should be provided (primary or metastatic).
8. Patients must have measurable lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
9. ECOG performance score 0 or 1.
10. Prior anti-tumor treatment-related AEs (NCI CTCAE v5.0 Criteria) have recovered to ≤ Grade 1 (except alopecia, non-clinically significant or asymptomatic laboratory abnormalities).
11. No severe cardiac dysfunction with left ventricular ejection fraction (LVEF) ≥ 50%.
12. Organ function must meet the basic requirements.
13. Coagulation function must meet the basic requirements.
14. Patients of childbearing potential must take effective contraceptive measures during the treatment and for 6 months after the last dose of treatment.

Exclusion Criteria:

1. History of hypersensitivity to any component of MRG002 or history of hypersensitivity of ≥ Grade 3 to trastuzumab.
2. Received radiotherapy, chemotherapy, biotherapy, immunotherapy, or other anti-tumor drugs within 4 weeks prior to the first dose MRG002 treatment.
3. Patients with clinical symptoms such as pleural, abdominal or pericardial effusion requiring puncture drainage.
4. Patients with central nervous system (CNS) metastasis and/or neoplastic meningitis.
5. Any severe or uncontrolled systemic diseases.
6. Patients with poorly controlled heart diseases.
7. Evidence of active infections, including but not limited to Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV) infection.
8. History of other primary malignancies.
9. History of interstitial pneumonia, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, etc.
10. Peripheral neuropathy greater than Grade 1.
11. History of cirrhosis (decompensated cirrhosis Child-Pugh class B and C).
12. Patients with active autoimmune disease or a history of autoimmune disease, who are using immunosuppressive agents, or systemic hormone therapy and still receiving within 2 weeks prior to enrollment.
13. Received anti-tumor vaccine treatment 4 weeks prior to the first dose or planning to participate in anti-tumor vaccine trials.
14. Female patents with a positive serum pregnancy test or who are breast-feeding or who do not agree to take adequate contraceptive measures during the treatment and for 6 months after the last dose of study treatment.
15. Other conditions inappropriate for participation in this clinical trial, at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by Independent Review Committee (IRC) | Baseline to study completion, up to 12 months
  ORR is defined as the percentage of patients with complete response (CR) and partial response (PR) as assessed by Independent Review Committee (IRC) according to RECIST v1.1.

SECONDARY OUTCOMES:
ORR by Investigator | Baseline to study completion, up to 12 months
  ORR is defined as the percentage of patients with CR and PR as assessed by Investigator according to RECIST v1.1.
Duration of Response (DoR) | Baseline to study completion, up to 12 months
  DOR is defined as the time from first documented objective response to the first onset of tumor progression or death of any cause.
Time to Response (TTR) | Baseline to study completion, up to 12 months
  TTR is defined as the duration from the start of treatment to the first onset of CR or PR in tumor evaluation.
Disease Control Rate (DCR) | Baseline to study completion, up to 12 months
  DCR is defined as the percentage of patients who achieve CR, PR, and stable disease (SD) after treatment.
Progression Free Survival (PFS) | Baseline to study completion, up to 12 months
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Overall Survival (OS) | Baseline to study completion, up to 12 months
  OS is defined as the duration from the start of treatment to death of any cause.
Adverse Events (AEs) | Baseline to 30 days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
Pharmacokinetics (PK) Parameter of MRG002: concentration-time curve | Baseline to 30 days after the last dose of study treatment
  Concentration-time curve will be depicted based on pharmacokinetics concentration set (PKCS).
Incidence of anti-drug antibody (ADA) | Baseline to 30 days after the last dose of study treatment
  The incidence of ADA analysis will be summarized for all patients who received at least one cycle study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (36):
- China (36):
  - Anhui provincial Cancer Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing hospital, Beijing, Beijing Municipality
  - Beijing Chao-Yang Hospital，Capital Medical University, Beijing, Beijing Municipality
  - The Fifth Medical Center of the PLA, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Army Medical Center of PLA, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - SUN Yat-sen university Cancer center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - ShenZhen Luohu People's Hospital, Shenzhen, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Haerbin medical university cancer hospital, Haerbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union hospital tongji medical college huazhong univerity ofscience and technology, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - Xiangya hospital central south university, Changsha, Hunan
  - The Affiliated Cancer Hospital of Xiangya School of Medicine(Hunan Cancer Hospital ), Changsha, Hunan
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - JiLinGuoWen Hospital, Siping, Jilin
  - Liaoning Cancer hospital, Shenyang, Liaoning
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Rui jin hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Xi'an Jiaotong University, Xian, Shanxi
  - Sichuan provincial people's hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The second Affiliated Hospital Zhejiang University School of Medical, Hangzhou, Zhejiang
  - Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang
  - The 1'Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No